CLINICAL TRIAL: NCT02018640
Title: Biomarker Feedback to Motivate Tobacco Cessation in Pregnant ALaska Native Women: Phase 2
Acronym: MAW Phase 2
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Alaska Native Tribal Health Consortium (Other); University of California, San Francisco (Other); University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Other Study IDs: 11-001144 Phase 2; U54CA153605 (NIH)
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cancer; Tobacco Use; Pregnancy
Keywords: cancer; tobacco use; pregnancy
MeSH Terms: conditions — Neoplasms; Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Use of tobacco is very high among Alaska Native pregnant women. The investigators are conducting a three phase study. The first study is nearly completed and involved measuring biomarkers of tobacco exposure in mothers and infants. The second phase of the research is a qualitative study to translate the biomarker findings to an intervention.

DETAILED DESCRIPTION:
Developing effective tobacco cessation interventions during pregnancy for American Indian and Alaska Native people is a national priority and will contribute to the U.S. public health objective of reducing tobacco-related cancer health disparities. The proposed project builds on our successful partnership with the Alaska Native community and previous work with Alaska Native pregnant women. We propose to develop and test a novel biomarker feedback intervention relating cotinine levels in the urine of pregnant women with the woman and infant's likely exposure to the tobacco specific nitrosamine and carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone) (NNK). This 5-year project will be conducted in three phases. In Phase 1 we utilized a non-randomized, clinical observational trial to examine biomarkers of nicotine and carcinogen exposure (urine cotinine and total NNAL [a metabolite of NNK], respectively) among maternal-infant pairs with assessments conducted during pregnancy and at delivery. In Phase 2, we will obtain qualitative feedback on the findings from Phase 1 through individual interviews conducted with women who use tobacco and a confidant (partner/friend/relative) they have identified to develop the biomarker feedback intervention messages. Phase 3 will consist of a formative evaluation of the biomarker feedback intervention with pregnant women using a two-group randomized design to assess the intervention's feasibility and acceptability, and the biochemically confirmed abstinence rate at the end of pregnancy. All phases of the project will be guided by a Community Advisory Committee. Each phase is an important step to advance our understanding of the potential for biomarker feedback as a strategy to help Alaska Native pregnant women quit tobacco use. The potential reach of the intervention is significant from a public health perspective as over 600 tobacco users deliver each year at the Alaska Native Medical Center in Anchorage where the proposed project will take place. Developing effective interventions for tobacco cessation during pregnancy is important to reduce adverse health consequences for the mother and neonate and future risk of tobacco-caused cancers.

ELIGIBILITY:
Inclusion Criteria:

To be eligible the woman must:

1. be Alaska Native
2. be aged 18 years of age or older
3. provide written informed consent
4. have participated in Phase 1 of the research or is currently pregnant (<= 24 weeks gestation)
5. have used any tobacco product at least once in the past 7 days (cigarettes or both cigarettes/ST)

To be eligible the confidant (he/she) must:

1. be referred by the woman participant
2. be aged 18 years of age or older
3. provide written informed consent

Exclusion Criteria:

1. does not provide written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Alaska Native women and their confidants
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
receptivity to cancer risk messages | baseline
  interview of participant reactions to biomarker findings

SECONDARY OUTCOMES:
confidant perceptions of cancer risk information | baseline
  interview of family members, friends, relatives

CONTACTS AND LOCATIONS:
Locations (1):
- Alaska Native Tribal Health Consortium, Anchorage, Alaska, United States